CLINICAL TRIAL: NCT02664636
Title: Pilot Study on the Development of Cortical Reorganization Models for Motor Areas and Inter-hemispheric Equilibrium in the Post-stroke Early Recovery Phase Evaluated by Functional Near-infrared Spectroscopy (fNIRS)
Brief Title: Cortical Reorganization Models for Motor Areas and Inter-hemispheric Equilibrium Post-stroke: a Pilot Study
Acronym: ERASM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2015/JF-02; 2015-A01624-45 (Other: ANSM)
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2016-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Experimental): The study population consists of patients 20 and 75 years of age who have had a supra-tentorial ischemic or hemorrhagic stroke. The study covers consulting or hospitalized patients at the neurological rehabilitation service (NHS) of Grau du Roi Medical Center, part of the Nîmes University Hospital. Most patients originate from a 2-4 week stay in the neurological acute care, cardiac or polyvalent departments of the University Hospitals of Montpellier or Nîmes.
  Intervention: Physiotherapy
  Intervention: Occupational therapy
  Intervention: Functional near-infrared spectroscopy
  Interventions: Procedure: Physiotherapy; Procedure: Occupational therapy; Procedure: Functional near-infrared spectroscopy

INTERVENTIONS:
Procedure: Physiotherapy — Physiotherapy regimen (days 0 to 60): orthopedic maintenance, work on trunk balance, sensorimotor techniques for restoration of motor skills, exercises for standing balance and walking. Sessions last 30 to 60 minutes depending on the fatigue of the subject and the level of recovery. They occur as daily sessions during the first two weeks and then two sessions / day.
  This is part of routine care.
Procedure: Occupational therapy — Occupational Therapy (days 0 to 60): Orthopaedic maintenance, exercises for sitting and standing balance, sensorimotor techniques for the restoration of motor skills, grip exercises. Sessions last 30 to 60 minutes depending on the fatigue of the subject and the level of recovery. 1 session is performed per day.
  This is part of routine care.
Procedure: Functional near-infrared spectroscopy — During the therapy protocol, cortical activation measures using the fNIRS method will be conducted every 15 days (at Day0, Day 15, Day 30, Day 45 and Day 60 for 5 sessions in total) at the technical platform of the Grau du Roi physical therapy centre, during the completion of a standardized motor task (maintaining a level of force) using the healthy upper limb and the paretic upper limb.
  Other Names: fNIRS

SUMMARY:
The main objective is to develop models for the cortical reorganization of motor areas and inter-hemispheric equilibrium in the early phase of post stroke recovery evaluated by the fNIRS technique from day 0 to day 60 (day 0 being the day of inclusion in the study) and to correlate the latter with the early phases of motor recovery over the same period, as measured by the test Fugl-Meyer.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To evaluate changes in functional outcomes (Box and Blocks Test and NineHolePeg Test from Day 0 to Day 60.

B- To evaluate changes in autonomy (Barthel Index) from Day 0 to Day 60.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has had a first ischemic or haemorrhagic supra-tentorial stroke within the 2 to 4 weeks preceding inclusion

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient presents with a severe cognitive disorder
* The patient has severe aphasia with a Boston Diagnostic Aphasia Examination (BDAE) scale score strictly less than 2
* The patient has heminegligence with a bells test > 6 on the left.
* The patient presents with limited amplitude in the paretic upper limb (shoulder abduction <60°, elbow flexion > 30° or dorsal wrist flexion <20°).
* Imbalanced/uncontrolled epilepsy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Near-infrared spectroscopy signal analysis: the average amplitude of cortical activation | Day 0
Near-infrared spectroscopy signal analysis: the average amplitude of cortical activation | Day 15
Near-infrared spectroscopy signal analysis: the average amplitude of cortical activation | Day 30
Near-infrared spectroscopy signal analysis: the average amplitude of cortical activation | Day 45
Near-infrared spectroscopy signal analysis: the average amplitude of cortical activation | Day 60
Near-infrared spectroscopy signal analysis: the amplitude peak | Day 0
Near-infrared spectroscopy signal analysis: the amplitude peak | Day 15
Near-infrared spectroscopy signal analysis: the amplitude peak | Day 30
Near-infrared spectroscopy signal analysis: the amplitude peak | Day 45
Near-infrared spectroscopy signal analysis: the amplitude peak | Day 60
Near-infrared spectroscopy signal analysis: the time required to reach the peak | Day 0
Near-infrared spectroscopy signal analysis: the time required to reach the peak | Day 15
Near-infrared spectroscopy signal analysis: the time required to reach the peak | Day 30
Near-infrared spectroscopy signal analysis: the time required to reach the peak | Day 45
Near-infrared spectroscopy signal analysis: the time required to reach the peak | Day 60
Near-infrared spectroscopy signal analysis: the laterality index | Day 0
Near-infrared spectroscopy signal analysis: the laterality index | Day 15
Near-infrared spectroscopy signal analysis: the laterality index | Day 30
Near-infrared spectroscopy signal analysis: the laterality index | Day 45
Near-infrared spectroscopy signal analysis: the laterality index | Day 60
Voluntary force: the target error which measures the difference between the average of the force developed by the arm and target strength | Day 0
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: the target error which measures the difference between the average of the force developed by the arm and target strength | Day 15
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: the target error which measures the difference between the average of the force developed by the arm and target strength | Day 30
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: the target error which measures the difference between the average of the force developed by the arm and target strength | Day 45
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: the target error which measures the difference between the average of the force developed by the arm and target strength | Day 60
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: average | Day 0
  Voluntary force refers to the force applied during motricity tasks. "Average" refers to the sum of measures weighted by the number of measures.
Voluntary force: average | Day 15
  Voluntary force refers to the force applied during motricity tasks. "Average" refers to the sum of measures weighted by the number of measures.
Voluntary force: average | Day 30
  Voluntary force refers to the force applied during motricity tasks. "Average" refers to the sum of measures weighted by the number of measures.
Voluntary force: average | Day 45
  Voluntary force refers to the force applied during motricity tasks. "Average" refers to the sum of measures weighted by the number of measures.
Voluntary force: average | Day 60
  Voluntary force refers to the force applied during motricity tasks. "Average" refers to the sum of measures weighted by the number of measures.
Voluntary force: coefficient of variation | Day 0
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: coefficient of variation | Day 15
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: coefficient of variation | Day 30
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: coefficient of variation | Day 45
  Voluntary force refers to the force applied during motricity tasks.
Voluntary force: coefficient of variation | Day 60
  Voluntary force refers to the force applied during motricity tasks.
Fugl-Meyer motricity score | Day 0
  The Fugl-Meyer motricity score includes evaluations of tone, strength and motor skills.
Fugl-Meyer motricity score | Day 15
  The Fugl-Meyer motricity score includes evaluations of tone, strength and motor skills.
Fugl-Meyer motricity score | Day 30
  The Fugl-Meyer motricity score includes evaluations of tone, strength and motor skills.
Fugl-Meyer motricity score | Day 45
  The Fugl-Meyer motricity score includes evaluations of tone, strength and motor skills.
Fugl-Meyer motricity score | Day 60
  The Fugl-Meyer motricity score includes evaluations of tone, strength and motor skills.

SECONDARY OUTCOMES:
The Box and Block test: The score is the number of blocks transferred in one minute. | Day 0
The Box and Block test: The score is the number of blocks transferred in one minute. | Day 60
The Nine Hole Peg Test: The score is the total time to complete the task. | Day 0
The Nine Hole Peg Test: The score is the total time to complete the task. | Day 60
The Barthell test for autonomy | Day 0
The Barthell test for autonomy | Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Froger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Nîmes - Hôpital Universitaire de Réadaptation du Grau du Roi, Le Grau-du-Roi
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delorme M, Vergotte G, Perrey S, Froger J, Laffont I. Time course of sensorimotor cortex reorganization during upper extremity task accompanying motor recovery early after stroke: An fNIRS study. Restor Neurol Neurosci. 2019;37(3):207-218. doi: 10.3233/RNN-180877. PMID 31227675